CLINICAL TRIAL: NCT03927287
Title: An "Old" Biomarker That Can Learn New Tricks: Prognostic Role of Free Psa Ratio at Biochemical Recurrence After Radical Treatments for Prostate Cancer
Brief Title: Prognostic Role of Free Psa Ratio at Biochemical Recurrence After Radical Treatments for Prostate Cancer
Acronym: FPSAR
Status: Completed | Type: Observational
Sponsor: Rabin Medical Center (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Principal Investigator, Hanan Goldberg, Principal Investigator, University of Toronto
Other Study IDs: 17-5498
Record Dates: First submitted 2019-04-19; First posted 2019-04-25 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Metastasis; Castration-resistant Prostate Cancer; Death
MeSH Terms: conditions — Neoplasm Metastasis; Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Radical prostatectomy (RP cohort): Our institutional prostate cancer database was queried for all patients between 2000-2017 who had a biochemical recurrence (BCR) after radical prostatectomy (RP) (Total PSA>=0.2 ng/ml) and had at least one post-BCR free PSA ratio (FPSAR) blood test (RP cohort). FPSAR ascertainments were performed incidentally or reflexively (e.g. PSA in the range of 4-10 ng/ml, as per Institutional policy). If multiple FPSAR tests were performed, only the first FPSAR test was analyzed. otal PSA and Free PSA data was performed with the Abbott Architect analytical platform, according to the instructions of the manufacturer.
- Radiotherapy cohort: Our institutional database was queried or all patients between 2000-2017 who had a rising PSA after radiotherapy (RT) for intermediate- and high-risk prostate cancer, and at least one post-treatment free PSA ratio (FPSAR) blood test (RT cohort). As in the RP cohort, FPSAR was performed either incidentally or reflexively, and the first FPSAR test was used for the analyses. Total PSA and Free PSA data was performed with the Abbott Architect analytical platform, according to the instructions of the manufacturer.
- Biobank surgical cohort: To validate our findings in the two retrospective cohorts (RP and RT), we analyzed a third cohort of prospectively collected biobank specimens of patients who underwent RP and developed biochemical recurrence(Biobank cohort). The retrieved samples were batched and tested for FPSAR levels to determine the results in lower PSA ranges and also to account for intrinsic analyte measurements variability in the retrospective cohorts. For his cohort we used the Roche Elecsys analytical platform, according to the instructions of the manufacturer.
  Interventions: Diagnostic Test: Free PSA ratio test in patients after definitive treatment for localized prostate cancer

INTERVENTIONS:
Diagnostic Test: Free PSA ratio test in patients after definitive treatment for localized prostate cancer — Free PSA ratio blood test done on biobank samples of patients after radical prostatectomy who developed biochemical recurrence.
  Groups: Biobank surgical cohort

SUMMARY:
Measurement of Free PSA ratio in patients after definitive radical treatment for prostate cancer, and assessment of whether post-treatment free PSA ratio can function as a biomarker for advanced disease in prostate cancer patients.

DETAILED DESCRIPTION:
Prostatic specific antigen (PSA) circulates mostly in complex with protease inhibitors, but 10-30% circulates as inactive free-PSA (FPSA). In patients with prostate cancer (PCa), pretreatment FPSA is lower and used to risk-stratify patients for biopsy. However, posttreatment FPSA ratio (FPSAR) is rarely quantified, with an unexplored clinical value.

Methods The institutional database was queried to identify patients following radical prostatectomy (RP cohort) or radiotherapy (RT cohort) between 2000 and 2017. For validation, the investigators identified an independent prospective cohort with biochemical recurrence (BCR) after RP, using biobank samples (biobank cohort). All patients had at least one posttreatment FPSAR test. Kaplan-Meier (KM) method was used to compare the metastasis-free (MFS), castration-resistant PCa (CRPC)-free, and cancer-specific-survival (CSS) rates. Multivariable Cox models determined the association between posttreatment FPSAR, metastases, and CRPC.

ELIGIBILITY:
Inclusion Criteria:

For the two retrospective cohorts:

1. All patients that older than 18 treated for localized adenocarcinoma of the prostate between 2000 and 2017 with either radical prostatectomy or radiotherapy
2. All treated patients had a rising post-treatment PSA, with at least one post-treatment free PSA blood test.

For the biobank validation cohort:

1. All patients treated with radical prostatectomy for localized prostate cancer between 2000 and 2017 who had biobank samples taken when developing biochemical recurrence.

Exclusion Criteria:

1. Patients that were younger than 18,
2. Patients with prostate cancer other than adenocarcinoma, such as small cell and neuroendocrine cancer
3. Patients with prostate adenocarcinoma that did not develop biochemical recurrence.
4. In the retrospective cohorts - patients that did not have at least one post-treatment free PSA blood test.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Must be men with prostate cancer
Study Population: All patients in Princess Margaret Cancer treated for localized adenocarcinoma of the prostate between 2000 and 2017 with either radical prostatectomy or radiotherapy with a rising post-treatment PSA, who had at least one post-treatment free PSA blood test.
Sampling Method: Non-Probability Sample
Enrollment: 822 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2019-04-10 (Actual)

PRIMARY OUTCOMES:
Metastasis free survival | From date of diagnosis to date of Metastasis development, assessed up to 200 months
  Rate of Metastasis correlated to the first post-treatment free PSA ratio

SECONDARY OUTCOMES:
Castrate resistant prostate cancer (CRPC) free survival | From date of Diagnosis to date of CRPC development, assessed up to 200 months
  Rate of CRPC correlated to the first post-treatment free PSA ratio
Cancer specific survival | From date of diagnosis to date of cancer specific death, assessed up to 200 months
  Rate of Cancer specific survival correlated to the first post-treatment free PSA ratio

CONTACTS AND LOCATIONS:
Overall Officials: Neil Fleshner, MD, MPH, Study Director — Princess Margaret Hospital, University Health Network
Locations (1):
- Princess Margaret Cancer Center, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goldberg H, Glicksman R, Woon D, Hoffman A, Shaikh H, Chandrasekar T, Klaassen Z, Wallis CJD, Ahmad AE, Sanmamed-Salgado N, Qu X, Moraes FY, Diamandis EP, Berlin A, Fleshner NE. Can post-treatment free PSA ratio be used to predict adverse outcomes in recurrent prostate cancer? BJU Int. 2021 Jun;127(6):654-664. doi: 10.1111/bju.15236. Epub 2020 Sep 26. PMID 32926761